CLINICAL TRIAL: NCT03847844
Title: Cytopeutics® Umbilical Cord Mesenchymal Stem Cells (Cyto-MSC) for Patients With Grade II -IV Acute Graft-Versus-Host Disease: A Phase I/II Clinical Study
Brief Title: UCMSCs as Front-line Approach of Treatment for Patients With aGVHD
Acronym: GVHD Cyto-MSC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cytopeutics Sdn. Bhd. (Industry)
Collaborators: Universiti Tunku Abdul Rahman (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: POD0030/CP/R
Record Dates: First submitted 2019-02-14; First posted 2019-02-20 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Acute-graft-versus-host Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Cyto-MSC (5 million UCMSCs per kg bodyweight) and standard treatment
  Interventions: Biological: Umbilical cord derived mesenchymal stem cell
- Group B (Placebo Comparator): Placebo (normal saline) and standard treatment
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Umbilical cord derived mesenchymal stem cell — Umbilical cord derived mesenchymal stem cell
  Other Names: Cyto-MSC
  Arms: Group A
Other: Placebo — Normal saline
  Arms: Group B

SUMMARY:
Background: Graft-versus-host disease (GVHD) is a devastating complication following allogeneic hematopoietic stem cell transplantation (HSCT) mediated by stimulation of antigen presenting cells (APCs) which leads to donor T-lymphocytes activation and target tissue destruction, particularly affecting the skin, gastrointestinal tract, and liver in acute setting. In recent years, researchers have discovered that the application of mesenchymal stromal cells (MSCs) as salvage treatment among steroid refractory GVHD patients improves outcomes without long-term risk association. On the other hand, the use of MSCs concurrently with steroids as front-line treatment for acute GVHD has yet to be researched on. The investigators hypothesize that this approach, as the MSCs will be administered at earlier stage of the disease, will increase survival rate and reduce mortality among aGVHD patients.

Objective: In this study, the investigators aim to determine the efficacy and safety of allogeneic infusion of Cytopeutics® umbilical cord-derived mesenchymal stromal cells (Cyto-MSC) in combination of standard corticosteroid therapy as front-line approach for treatment of grade II-IV acute GVHD patients.

Study design: This is a phase I/II clinical study involving patients who underwent an allogeneic HSCT for malignant or non malignant haematological disorders and developed grade II-IV acute GVHD. A total of 40 eligible patients will be recruited in this study.

For Phase I open labelled study, 5 eligible patients will be recruited to receive Cyto-MSC (5 million UC-MSCs per kg bodyweight) and standard treatment. Meanwhile, for Phase II double blinded placebo controlled study, another 35 eligible patients will be recruited and randomized into 2 study groups where 15 patients will be assigned into Group A to receive Cyto-MSC (5 million UCMSCs per kg bodyweight) and standard treatment, meanwhile another 20 patients will be assigned into Group B to receive Placebo and standard treatment.

Cyto-MSC or Placebo will be administered at Day 1 and Day 4. Another infusion of Cyto-MSC or Placebo will be given at Day 7 if the patient shows no or partial response based on GvHD grading criteria. All patients will be assessed up until 6 months follow-up which include medical history, clinical and physical evaluations, pathology investigations, biomarkers and immune cell subsets analysis, as well as quality of life questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Patient age 16 and above
* Patient who has undergone an allogeneic haematopoietic stem cell transplantation (HSCT) receiving allograft either from HLA-matched related donor (MRD), HLA-matched unrelated donor (MUD), Unrelated Cord Blood (UCB) or Haploidentical donor and developed grade II-IV acute graft versus host disease (acute GVHD) involving the skin, GI tract and/or liver based on 1994 Consensus Conference on Acute GVHD Grading
* Patient and/or parent(s) or legal guardian(s) and assent form signed informed consent. Assent form will be obtained for patients aged less than 18 years. Investigators will obtain the permission of the parents or guardians for the participation of the minor in the research, and to solicit assent from the minor

Exclusion Criteria:

* Patient who has enrolled in another investigational drug trial or stem cell related trial or has completed the aforesaid within (3) months
* Patient with HIV or syphilis (Patient should be screened for HIV and VDRL up to 6 months prior to study start)
* Patient with Hepatitis B (HBV) or Hepatitis C (HCV). All patients must be screened for HBV and HCV up to 6 months prior to study start using the routine hepatitis virus laboratory. Patients who are positive for HBsAg or HBcAb will be eligible if they are negative for HBV-DNA, these patients should receive prophylactic antiviral therapy. Patients who are positive for anti-HCV antibody will be eligible if they are negative for HCV-RNA
* Patient has creatinine clearance of ≤50mL/min or creatinine is ≥200 µmol/L
* Patient had undergone or on other immune-modulatory treatments such as interferon or Thalidomide over the last 12 months
* Patient with progressive underlying disease or not in complete remission (CR) at the time of transplant
* Any other severe co-morbidities which the doctor deems as a contraindication to cell therapy
* Adults under law protection or without ability to consent
* The patient has previous history or on-going psychiatric illness
* Patient has received an HSCT transplant for a solid tumor disease
* Patient has a known hypersensitivity to dimethyl sulfoxide (DMSO)
* Patient is a female who is pregnant, lactating, or is planning a pregnancy during study participation, or in the follow-up period

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2023-07-18 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Rate of Complete Response (CR) at Day 28 | 28 days
Rate of Partial Response (PR) at Day 28 | 28 days
Rate of PR and CR at Day 14 | 14 days
Percentage of patient requiring MMF rescue during treatment | 6 months
Rate of long term complication incidence | 6 months
Rate of chronic clinical response incidence | 6 months

SECONDARY OUTCOMES:
Overall survival (OS) rate at 3 months | 3 months
Correlation between response to Cyto-MSC at Day 14 and Day 28 to survival at 90 days | 90 days
Relapse-free survival at 3 months | 3 months
Disease relapse at 3 months | 3 months
Incidence of infection | 6 months
Incidence of CMV reactivation | 6 months
Measurement quality of life of cancer patients by using EORTC QLQ-C30 questionnaire | 6 months
  The final score ranges from 0 (better outcome) to 126 (worse outcome)
Measurement quality of life in bone marrow transplantation by using FACT-BMT questionnaire | 6 months
  The final score ranges from 0 (better outcome) to 164 (worse outcome)
Measurement of health-related quality of life in children and young people by using PEDsQL questionnaire (patients age less than 18 years old) | 6 months
  The final score ranges from 0 (better outcome) to 92 (worse outcome)
Measurement of generic health status among patients by using EQ-5D questionnaire | 6 months
  The final score ranges from 0 (better outcome) to 100 (worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Sen Mui Tan, Principal Investigator — Hospital Ampang
Locations (1):
- Hospital Ampang, Ampang, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No